CLINICAL TRIAL: NCT01028742
Title: Posttraumatic Hypopituitarism - Incidence, Predictors and Test Validity
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Christina Klose, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: H-B-2008-122
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury; Hypopituitarism
Keywords: Traumatic brain injury; Hypopituitarism; Incidence
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypopituitarism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to estimate the incidence of posttraumatic hypopituitarism, and to identify predisposing factors in order to establish a rational responsible socioeconomic screening program.

ELIGIBILITY:
Inclusion Criteria:

* International Classification of Diseases (ICD) 10 code S06.0-06.9
* Age 18 - 65 years at time of traumatic brain injury
* Duration of hospitalization > 24 hours.

Exclusion Criteria:

* Known pituitary disease
* Clinically significant liver or renal disease
* Breast-feeding
* Pregnancy
* Alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised with a traumatic brain injury at any danish hospital between 01.01.2008 - 31.12.2008
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hypopituitarism | 5 years

SECONDARY OUTCOMES:
Quality of life | 5 years
Fatigue | 5 years
Hypopituitary specific symptoms | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD, Study Chair — Dept of Endocrinology, Rigshospitalet

REFERENCES:
- [Derived] Klose M, Stochholm K, Janukonyte J, Christensen LL, Cohen AS, Wagner A, Laurberg P, Christiansen JS, Andersen M, Feldt-Rasmussen U. Patient reported outcome in posttraumatic pituitary deficiency: results from The Danish National Study on posttraumatic hypopituitarism. Eur J Endocrinol. 2015 Jun;172(6):753-62. doi: 10.1530/EJE-14-1069. Epub 2015 Mar 12. PMID 25766045